CLINICAL TRIAL: NCT01632774
Title: Analysis of Risk Factors for Death After Blunt Traumatic Rupture of the Thoracic Aorta
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: TAR
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Aortic Rupture
MeSH Terms: conditions — Aortic Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aortic injuries after blunt thoracic trauma are compared to the great incidence of accidents relatively rare, but potentially serious leading to death at scene in most of the cases. The study was undertaken to delineate mortality and its risk factors on three different levels (pre-hospital, in-hospital and overall). Between 1990 and 2003, all consecutive patients and victims with traumatic aortic rupture were retrospectively analyzed by reviewing hospital and autopsy records.

DETAILED DESCRIPTION:
During the study period of 14 years (January 1990 to December 2003), all consecutive cases with traumatic rupture of the thoracic aorta being reported in the greater area of Zurich with about one million inhabitants were included in the present study. Related to the final outcome, patient data were drawn either from medical reports from the University Hospital of Zurich, which is a tertiary care teaching hospital and level I trauma center for the eastern part of Switzerland, or from autopsy reports from the Institute of Forensic Medicine of the University of Zurich, respectively. The latter group includes all patients, who died on the scene, in a assigning primary care hospital or on the way to the University Hospital of Zurich. In Switzerland, the criteria used for performing a full autopsy after a blunt traumatic death include all cases in which the events leading to the death are unclear or in which the cause of death is the result of suicide or extrinsic harm. Both, deaths at the scene and in-hospital deaths were included in the study.

ELIGIBILITY:
Inclusion criteria:

* During the study period of 14 years (January 1990 to December 2003), all consecutive cases with traumatic rupture of the thoracic aorta being reported in the greater area of Zurich with about one million inhabitants were included in the present study

Exclusion criteria:

* Non-traumatic aortic rupture
* Non-traumatic aortic dissection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients Patients who died at the scene
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 1990-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Division of Internal Medicine
Locations (1):
- University Hospital Zurich, Division of Internal Medicine, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Franzen D, Genoni M. Analysis of risk factors for death after blunt traumatic rupture of the thoracic aorta. Emerg Med J. 2015 Feb;32(2):124-9. doi: 10.1136/emermed-2013-202639. Epub 2013 Sep 4. PMID 24005640